CLINICAL TRIAL: NCT02402140
Title: A Prospective Randomized Trial Investigating the Influence of Pharmaceutical Care on the Intraindividual Variability of Tacrolimus Concentrations Early After Kidney Transplant.
Brief Title: Influence of Pharmaceutical Care on the Intraindividual Variability of Tacrolimus Concentrations
Acronym: PharmCare
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital do Rim e Hipertensão (Other)
Responsible Party: Principal Investigator, Adrieli Barros Bessa, Pharmacist, Hospital do Rim e Hipertensão
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: Hospital do Rim
Record Dates: First submitted 2015-03-06; First posted 2015-03-30 (Estimated); Last update posted 2015-11-03 (Estimated); Status verified 2015-10

CONDITIONS: Renal Transplant Graft Failure
Keywords: tacrolimus blood concentration; pharmaceutical intervention; intrasubject variability

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 with pharmaceutical intervention (Experimental): Patients allocated to group 1 with pharmaceutical intervention received instructions on the proper use of immunosuppressants as dosage, frequency and administration schedules, importance of immunosuppressive drugs and the risk of rejection.
  No more interventions were applied.
  Interventions: Other: Pharmaceutical Intervention
- 2 without pharmaceutical intervention (No Intervention): Standard following of the Hospital do Rim, without pharmaceutical intervention. This group was just followed by the nurses of the hospital, but without a standardized intervention.
  It was not a intervention, it was the control group

INTERVENTIONS:
Other: Pharmaceutical Intervention — Patients allocated to group 1, with pharmaceutical intervention, received instructions on the proper use of immunosuppressants as doses, frequency, importance, schedules on the following days 3, 5, 7, 10, 14, 21, 28, 60 and 90 after kidney transplant. Teaching materials were designed to assist in the pharmaceutical guidelines that understood the importance of immunosuppressive drugs, the risk of rejection, the schedules and the most appropriate way for the administration. In addition to these guidelines, pharmacists helped patients in filling out the patient diary. This diary contains all the medications that the patient administers and encourages them to write down daily doses in order to remind them. This was a standardized pharmacist intervention.
  Arms: 1 with pharmaceutical intervention

SUMMARY:
Primary end-point

The primary end-point was the influence of pharmaceutical intervention in tacrolimus intra-subject variability during the first 3 months after kidney transplant. Coefficients of variation were calculated from the average of dose-corrected tacrolimus blood concentration(CV= Standard Deviation (SD) x 100/mean) of study visits day 10, 14, 21, 30, 60 and 90 post kidney transplant.

Secondary end-points

1. Secondary outcomes included evaluate percentage of patients who achieved target levels of tacrolimus in day study visits 7, 10, 14, 21, 28, 60 e 90 days after kidney transplant;
2. Tacrolimus bioavailability profile during the period of 3 months,characterized by mean and standard deviation (SD) of dose corrected tacrolimus blood concentration(ng/ml/mg);
3. Assess patient adherence through validated questionnaire "Portuguese version of Basel Scale Adherence Rating Immunosuppressive Drugs (BAASIS) scale". It consists of a four-item questionnaire measuring nonadherence to immunosuppressives over the past four weeks. This questionnaire assesses omission of single doses or successive doses, timing deviations >2h and dose reductions. Responses are given on a six-point scale: never, once per month, every second week, every week, more than once per week and every day. Patients that answer different from "never" in any of the four questions are considered as nonadherent;
4. We evaluated renal function eGFR by Modification of Diet in Renal Disease (MDRD);
5. We evaluated Incidence of Infections;
6. We evaluated Treated acute rejection episodes;
7. We evaluated Death cases;
8. We evaluated Graft loss cases;
9. We evaluated Discontinuation of immunosuppressive treatment;
10. We evaluated Hospital readmissions.

Study Design

This was a single-center, prospective, randomized and controlled study to evaluate the influence of pharmaceutical intervention in tacrolimus intra-subject variability during the first 3 months after transplantation. The authors designed the protocol, acquired and maintained the data, and conducted the statistical analysis. The protocol was approved by an independent ethics committee. All subjects signed a written informed consent before enrollment and the study was conducted according to good clinical practices and declaration of Helsinki. This study was conducted at Hospital do Rim between February 2014 and December 2014, 128 randomized and were followed for 3 months after transplantation.

DETAILED DESCRIPTION:
Population

Inclusion criteria were patients who underwent renal transplantation aged ≥18 years old, who signed the informed consent, who underwent follow-up post transplant clinic at the Hospital do Rim for 3 months, receiving immunosuppressive drugs tacrolimus, prednisone and sodium mycophenolate or tacrolimus, azathioprine, and prednisone. Exclusion criteria were patients who underwent second kidney transplant, which did not follow the Hospital do Rim after transplant and who were participating in some other study with pharmaceutical intervention.

Randomization The randomization plan was carried out in blocks and stratified by immunosuppressive drugs tacrolimus, prednisone and mycophenolate sodium or tacrolimus, prednisone and azathioprine.

Opaque envelopes were made from a table of random numbers and they were open on the day of randomization to determine the group to which each patient was allocated group 1 with pharmaceutical intervention or group 2 without pharmaceutical intervention.

ELIGIBILITY:
Inclusion Criteria:

* patients who underwent renal transplantation aged ≥18 years old,
* who signed the informed consent,
* who underwent follow-up post transplant clinic at the Hospital do Rim for 3 months,
* receiving immunosuppressive drugs tacrolimus, prednisone and sodium mycophenolate or tacrolimus, azathioprine, and prednisone.

Exclusion Criteria:

* were patients who underwent second kidney transplant,
* which did not follow the Hospital do Rim after transplant and who were participating in some other study with pharmaceutical intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2014-02; Primary Completion 2014-10 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
The primary end-point was the influence of pharmaceutical intervention in tacrolimus intra-subject variability during the first 3 months after kidney transplant. variability during the first 3 months after transplantation. | 3 months
  Coefficients of variation were calculated from the average of dose-corrected tacrolimus blood concentration(CV= SD x 100/mean) of study visits day 10, 14, 21, 30, 60 and 90 post kidney transplant.

SECONDARY OUTCOMES:
Assess patient adherence through validated questionnaire "Portuguese version of BAASIS scale (Basel Scale Adherence Rating Immunosuppressive Drugs)"; | 3 months
  It consists of a four-item questionnaire measuring nonadherence to immunosuppressives over the past four weeks. This questionnaire assesses omission of single doses or successive doses, timing deviations >2h and dose reductions. Responses are given on a six-point scale: never, once per month, every second week, every week, more than once per week and every day. Patients that answer different from "never" in any of the four questions are considered as nonadherent.
Secondary outcomes included evaluate percentage of patients who achieved target levels of tacrolimus in day study visits day 7, 10, 14, 21, 28, 60 e 90 post kidney transplant | 3 months
We also evaluated renal function (eGFR by MDRD formula) | 3 months
Tacrolimus bioavailability profile during the period of 3 months | 3 months
  Characterized by mean and standard deviation of dose corrected tacrolimus blood concentrations(ng/ml/mg)
We evaluated the incidence of Infections | 3 months
We evaluated treated acute rejection episodes | 3 months
We evaluated death cases | 3 months
We evaluated graft loss cases | 3 months
We evaluated discontinuation of immunosuppressive treatment | 3 months
We evaluated hospital readmissions. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Adrieli BA Bessa, Pharmacist, Principal Investigator — Hospital do Rim

REFERENCES:
- [Derived] Mellon L, Doyle F, Hickey A, Ward KD, de Freitas DG, McCormick PA, O'Connell O, Conlon P. Interventions for increasing immunosuppressant medication adherence in solid organ transplant recipients. Cochrane Database Syst Rev. 2022 Sep 12;9(9):CD012854. doi: 10.1002/14651858.CD012854.pub2. PMID 36094829